CLINICAL TRIAL: NCT04796103
Title: The Effectiveness of Prolotherapy (%5 Dextros) in the Treatment of Patients With Chondromalacia Patella: a Randomized Controlled Trial
Brief Title: The Effectiveness of Prolotherapy (%5 Dextros) in the Treatment of Patients With Chondromalacia Patella
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9
Record Dates: First submitted 2020-12-19; First posted 2021-03-12 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Chondromalacia Patellae
Keywords: prolotherapy; knee pain; ultrasound; exercise
MeSH Terms: conditions — Chondromalacia Patellae; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose Prolotherapy Group (Active Comparator): Patients diagnosed with chondromalacia patella
  Interventions: Procedure: Dextrose Prolotherapy; Procedure: Serum Physiological Group (placebo control group)
- Serum Physiological Group (Placebo Comparator): Patients diagnosed with chondromalacia patella
  Interventions: Procedure: Dextrose Prolotherapy; Procedure: Serum Physiological Group (placebo control group)

INTERVENTIONS:
Procedure: Dextrose Prolotherapy — In the patients in the prolotherapy injection group, at the 1st, 4th and 7th weeks, the insertion points of the ligaments and tendons that are sensitive with pressure around the knee (medial collateral ligament (2), lateral collateral ligament (2), quadriceps tendon (1) and patellar tendon (1)) A total of 6 ml of 5% dextrose, 1 ml each, will be applied periarticularly. In addition, home exercise program will be given to this group.
Procedure: Serum Physiological Group (placebo control group) — In the patients in serum physiological injection group, at the 1st, 4th and 7th weeks, the insertion points of the ligaments and tendons that are sensitive with pressure around the knee (medial collateral ligament (2), lateral collateral ligament (2), quadriceps tendon (1) and patellar tendon (1)) A total of 6 ml of saline will be applied periarticularly. In addition, home exercise program will be given to this group.

SUMMARY:
Dextrose prolotherapy is a form of treatment in which hypertonic dextrose solution is used as a stimulant solution and regeneration is increased by stimulating the body's natural healing mechanisms after injection.

The aim of this study is to compare the dextrose prolotherapy applied with home exercise program and saline injections as a control group in patients who applied to our clinic with knee pain and diagnosed with chondromalacia patella, and to investigate the effectiveness of dextrose and saline on the job to determine the superiority of the injections to each other.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. 48 people who met the inclusion criteria were randomized into two groups of 24 people. The first group will be designated as Dextrose Prolotherapy Group and dextrose prolotherapy and exercise program will be applied to these patients. Patients in the second group will be designated as the Serum Physiological Group, and injections with saline and home exercise program will be applied in accordance with the prolotherapy protocol.Participants were evaluated with Visual Analogue Scale (VAS), Patello Femoral Pain Severity Scale (PFPSS), Kuala Patellofemoral Scoring System (KPSS) and Short Form 36 (SF-36).Knee cartilage thickness measurements and the presence of suprapatellar effusion of the participants whose evaluations are completed will be evaluated bilaterally by ultrasonography and the findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female / male aged> 18 years
* Diagnosis of chondromalacia patella after physical examination and imaging (direct radiography, MRI)
* Those whose symptoms persist> 3 months
* Does not have a disease that will prevent him from exercising
* Participation in the study voluntarily and regularly

Exclusion Criteria:

* Pregnant patients
* History of previous knee surgery
* Having received physical therapy from the knee area in the last 3 months
* Drug allergy
* Previous prolotherapy or any injection up to 3 months ago
* Those with pain reflected from waist or hip
* Patients with neuropathic pain
* Tumor, infectious, psychiatric illness, history of bleeding diathesis
* Having a trauma history in the last 6 months
* Those with systemic diseases such as diabetes, hepatitis, coagulopathy
* Those with cerebrovascular event disease in which bleeding continues actively
* Those who received NSAID treatment within the last week
* Patients with a BMI> 40
* Finding leg length difference

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Knee Pain | initial, 4th week 7th week 24th week pain change
  Severity of pain was assessed using the standard 10 cm VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end

SECONDARY OUTCOMES:
Patello Femoral Pain Intensity Scale | initial, 4th week 7th week 24th week pain change
  Patello Femoral Pain Intensity Scale to evaluate patients' pain in climbing / descending stairs, squatting, walking, jogging, sprinting, sports, sitting for 20 minutes with knees flexed at 90 °, standing on the knee, resting and resting after an activityStair climbing / descending, crouching, walking, jogging, sprinting, sports, sitting for 20 minutes with knees flexed at 90 °, standing on the knee, resting and resting after an activity, travel 10 cm as standard 0 "no pain" at one end, 10 At the other end it was rated as "excruciating pain" with a total score of 100.

OTHER OUTCOMES:
Kuala Patellofemoral Scoring System | initial, 4th week 7th week 24th week changes
  Kuala Patellofemoral Scoring System was used to determine the functional levels of the patients. Participants were evaluated over a minimum of 0 and a maximum of 100 points.
Short Form-36 (SF-36) | initial, 4th week 7th week 24th week changes
  Short Form (SF-36) was used to investigate the quality of life of the patients.The reliability and validity of the Turkish version of SF-36 has been demonstrated. SF-36 consists of 36 questions on eight different subscales including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy and fatigue, vitality, social functioning, role limitations due to emotional problems and general mental health. Each subscale of SF-36 is scored between 0 and 100, and higher scores show better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem KÖROĞLU, MD, Study Director — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Burak BAYIR, MD, Principal Investigator — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No